CLINICAL TRIAL: NCT00757445
Title: Treatment Results on Patients With Debridement and Prosthesis Retention in the Hip 1997-2007
Brief Title: Treatment Results on Patients With Debridement and Prosthesis Retention in the Hip
Status: Completed | Type: Observational
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Bjoern Waagsboe, Sorlandet Sykehus HF
Other Study IDs: Sorlandet Hospital HF
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Infection; Debridement With Prosthesis Retention
Keywords: Antibiotic therapy; Microbiological diagnosis
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study presents the investigators results on patients treated for infection in the implemented hip prosthesis. Debridement and prosthesis retention is the method, followed by antibiotic treatment. The investigators present treatment results, predisposing factors and microbiological data.

ELIGIBILITY:
Inclusion Criteria:

* Infection in prothesis in hip treated with debridement and prosthesis retention

Exclusion Criteria:

* Other technique

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with prosthesis infection in hip
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 1997-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bjoern Waagsboe, MD, Principal Investigator — Sorlandet Hospital HF
Locations (1):
- Sorlandet Hospital HF, Kristiansand, Agder, Norway